CLINICAL TRIAL: NCT04135677
Title: A Multi-center Randomized Controlled Study of High/Low-dosage Rivaroxaban Compared With DAPT After Left Atrial Appendage Occulsion in Patients With Non-valvular Atrial Fibrillation（ESCORT-AF Study(B)）
Brief Title: Clinical Outcomes Between Anticoagulation and DAPT Therapy in AF Patients Successfully Undergoing LAAO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DRXCZ
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Left Atrial Appendage Thrombosis; Thrombi; Stroke
MeSH Terms: conditions — Thrombosis; Stroke | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAPT group (Active Comparator): asprin 100mg qd together clopidogrel 75mg for 24 weeks
  Interventions: Drug: DAPT
- Anticoagulation group (Experimental): rivaroxaban 20mg qd for for 12 weeks and continued DAPT(asprin 100mg qd together clopidogrel 75mg) for 24 weeks
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Drug: Rivaroxaban 20mg Duration of treatment: 12 weeks(12 weeks for DAPT afterwards)
  Other Names: new oral anticoagulation
  Arms: Anticoagulation group
Drug: DAPT — Drug: Aspirin 100mg and clopidogrel 75mg Duration of treatment:24 weeks
  Other Names: dual antiplatelet therapy
  Arms: DAPT group

SUMMARY:
The objective of this study is to assess the efficacy and safety different dosage of rivaroxaban application versus dual antiplatelet therapy after successful closure of left atrial appendage using the LAMBRE device.

DETAILED DESCRIPTION:
Transcatheter left atrial appendage occlusion(LAAO) has emerged as an effective alternative for preventing thromboembolic events in patients with nonvalvular atrial fibrillation. The contemporary strategy for post-implantation antithrombotic medication therapy derived from several initial industrialized authoritative researches, demonstrated as 45 days for anticoagulation and prolonged DOAC for 6 months. In spite of the increasing experience of operators and arrival of new technologies, the rates of DRT still maintained. Therefore, whether altered medication therapy post-implantation attracted overwide attention. Nowadays, new oral anticoagulation such as rivaroxaban, dabigatran has evolved empirically and successively has been applied for days-weeks anticoagulation therapy following LAAO ,yet, the specific recommended dosage remained unclear.

Therefore, the objective of the study is to compare the effects of different dosage of rivaroxaban for short-term(12 weeks) anticoagulation therapy versus DAPT for post-LAAO anti-thrombotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Successful transcatheter LAAC using LAMBRE with COST criteria met by intra-procedural TEE and LAA angiography;
* Cha2ds2-Vasc2 score≥2 and or Has-bled score≥3(with contraindication or self-refusal to long-term administration of oral anticoagulants);
* Age18-85 years old;
* Life expectancy≥1 year;
* Written informed consent obtained;

Exclusion Criteria:

* • Prior history of cardiac surgery or with need for intervention in limited intervals;
* Intolerant of TEE or with clinical contraindications for TEE
* Detection of LAA/LA thrombus prior to the procedure;
* Anteroposterior diameter of LAA≥60mm according to TTE
* Impairment of renal function: eGFR≤15ml/min and/or creatinine level≥200μmol/L;
* Patients with hepatic disease that is associated with abnormal blood coagulation(cirrhosis: Child Pugh B an C);
* PLT ≤ 50*10^9/L;
* LVEF≤35% and/or NYHA≥IV；
* Allergies or contraindications to antiplatelet or anticoagulation therapy;
* At high risk of major bleedin(such as gastrointestinal ulcer at present or recently, malignant tumor with high risk of hemorrhage, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, angioaneurysms or major intraspinal or intracerebral vascular malformations, et al)
* Patients with requirement for anticoagulation therapy due to other diseases besides atrial fibrillation (such as after mechanical valve replacement, spontaneous or recurrent venous thromboembolism, etc.);
* Occurrence of severe pericardial tamponade, major hemorrhage and other life-threatening complications after left atrial appendage closure;
* Combined with other basic complications necessary to take drugs that may affect the effect of anticoagulation and antithrombotic regimen in this study(such as pyrrole antifungal agent, human acquired immunodeficiency virus (HIV) protease inhibitor, anti arrhythmia drug dronedarone, powerful cytochrome enzyme CYP3A4 inducer including rifampicin, phenytoin sodium, carbamazepine, phenobarbital, and other anticoagulants).
* Enrolled in other clinical studies in progress;
* Researches think that the patient is not suitable to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Primacy efficacy endpoint | 24 weeks after LAAC
  Number of participants with major adverse events(all-cause death, stroke/TIA, systematic embolism)
Primacy safety endpoint | 24 weeks after LAAC
  Number of participants with bleeding events(major or life-threatening)

SECONDARY OUTCOMES:
Device-related thrombosis | at 12-,24-week follow-up
  Number and rates of participants with DRT on TEE
Stroke | at 12,24-week follow-up
  Rates and distribution of participants withischemic and hemorrhagic stroke
Bleeding | at 12-,24-week follow-up
  Number and rates of participants with bleeding events in varying severity
Death | at 12-,24-week follow-up
  Number and rates of cardiovascular-related/not cardiovascular-related death
Re-hospitalization | at 12-,24-week follow-up
  Number and rates of participants indicated for re-hospitalization due to cardiovascular diseases
Composed endpoint | at 12-,24-week follow-up
  Number and rates of composed endpoints(DRT, rehospitalization for cardiovascular diseases and other primary endpoints)

CONTACTS AND LOCATIONS:
Overall Officials: JUNBO GE, PHD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan Univerisity, Shanghai, Shanghai Municipality, China